CLINICAL TRIAL: NCT06340828
Title: Washed Microbiota Transplantation Alleviates Diabetic Gastrointestinal Motility Disorders: an Efficacy and Safety Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-186-01
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Gastroparesis; Diabetic Gastropathy; Diabetic Gastroenteropathy; Diabetic Gastroparesis Associated With Type 2 Diabetes Mellitus
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Washing Microbiota Transplantation (WMT) group (Experimental): After assessing the general condition and gastrointestinal symptoms of the patients upon admission, consecutive days of washing microbiota transplantation were conducted. The administration time was 3 p.m., administered via a nasogastric tube at a dosage of 50 ml per administration. A follow-up appointment at the hospital was scheduled for week 12 post-treatment to reinforce the therapeutic effect with a second treatment, following the same timing, dosage, and administration route as the first treatment.
  Interventions: Other: Washing Microbiota Transplantation

INTERVENTIONS:
Other: Washing Microbiota Transplantation — Fecal samples from healthy adults were collected and underwent multiple centrifugations and filtrations to obtain a bacterial solution, which was then transplanted into the duodenum of patients via a nasogastric tube.
  Other Names: Fecal Microbiota Transplantation

SUMMARY:
The goal of this clinical trial is to learn about effectiveness and safety of washing microbiota transplantation in diabetic gastrointestinal motility disorders participant population. The main questions it aims to answer are:

* The risk factors of diabetic gastrointestinal motility disorders in routine clinical data or biochemical tests.
* The composition of gut microbiota in diabetic gastrointestinal motility disorders patients and potential pathogenic bacteria.
* The efficacy of washing microbiota transplantation in the clinical treatment of diabetic gastrointestinal motility disorders patients and potential factors that may influence treatment outcomes.
* The potential mechanisms of washing microbiota transplantation in treating diabetic gastrointestinal motility disorders patients.

Participants will be collected fasting venous blood and random stool samples before treatment and at week 12 post-treatment, conducting scale assessments before treatment and at weeks 1, 4, and 12 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes and diabetic gastrointestinal motility disorder.
* Glycated hemoglobin (HbA1c) < 11.0%.

Exclusion Criteria:

* Insulin dependent diabetes;
* Active infections, antibiotics-using, inflammatory bowel disease, irritable bowel syndrome, or other severe gastrointestinal organic disease;
* Severe diabetic complications;
* Thyroid disease, malignancies, severe cognitive impairment and mental disease;
* Alcohol or substance abuse;
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale | 0 days，weeks 1, 4, and 12 post-treatment
  Questionnaires，the minimum score is 0，and maximum is 45, and higher scores mean a worse outcome.
Gut Microbiome Sequencing | 0 days，weeks 12 post-treatment
  16S rRNA Sequencing

SECONDARY OUTCOMES:
Gastroparesis Cardinal Symptom Index | 0 days，weeks 1, 4, and 12 post-treatment
  Questionnaires，the minimum score is 0，and maximum is 45, and higher scores mean a worse outcome.
Composite Autonomic Symptom Score 31 | 0 days，weeks 1, 4, and 12 post-treatment
  Questionnaires，the minimum score is 0，and maximum is 75, and higher scores mean a worse outcome.
Gastrointestinal Motility | 0 days，weeks 12 post-treatment
  Neurophysiological Method
Heart Rate Variability | 0 days，weeks 12 post-treatment
  Neurophysiological Method
Serum Metabolites | 0 days，weeks 12 post-treatment
  Liquid chromatography-mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China